CLINICAL TRIAL: NCT06875310
Title: A Randomized, Double-Blind, Phase 3 Trial of Adagrasib Plus Pembrolizumab Plus Chemotherapy vs. Placebo Plus Pembrolizumab Plus Chemotherapy in Participants With Previously Untreated, Locally Advanced or Metastatic Non-squamous Non-small Cell Lung Cancer With KRAS G12C Mutation (KRYSTAL-4)
Brief Title: A Study of Adagrasib Plus Pembrolizumab Plus Chemotherapy vs. Placebo Plus Pembrolizumab Plus Chemotherapy in Participants With Previously Untreated Non-squamous Non-small Cell Lung Cancer With KRAS G12C Mutation (KRYSTAL-4)
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Mirati Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CA239-0004; CA2390004 (Other: Mirati Therapeutics Protocol ID)
Record Dates: First submitted 2025-03-07; First posted 2025-03-13 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: Immunotherapy; KRAS; KRAS G12C; Targeted therapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — adagrasib; pembrolizumab; Carboplatin; Pemetrexed; Cisplatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Adagrasib (Experimental)
  Interventions: Drug: Adagrasib; Drug: Pembrolizumab; Drug: Carboplatin; Drug: Pemetrexed; Drug: Cisplatin
- Placebo (Placebo Comparator)
  Interventions: Drug: Pembrolizumab; Drug: Carboplatin; Drug: Pemetrexed; Drug: Placebo; Drug: Cisplatin

INTERVENTIONS:
Drug: Adagrasib — Specified dose on specified days
  Other Names: BMS-986503; KRAZATI®
  Arms: Adagrasib
Drug: Pembrolizumab — Specified dose on specified days
  Other Names: KEYTRUDA®
Drug: Carboplatin — Specified dose on specified days
Drug: Pemetrexed — Specified dose on specified days
Drug: Placebo — Specified dose on specified days
  Arms: Placebo
Drug: Cisplatin — Specified dose on specified days

SUMMARY:
This is a trial to evaluate the efficacy, safety, and tolerability of adagrasib plus pembrolizumab plus platinum-doublet chemotherapy versus placebo plus pembrolizumab plus platinum-doublet chemotherapy in participants with previously untreated, locally advanced or metastatic NSCLC with KRAS G12C mutation

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed diagnosis of non-squamous NSCLC with evidence of KRAS G12C mutation via tumor sample and/or circulating tumor deoxyribonucleic acid (ctDNA).
* Locally advanced or metastatic disease.
* Measurable disease via computed tomography (CT) or magnetic resonance imaging (MRI) per RECIST v1.1 criteria of at least 1 lesion.
* No prior systemic anti-cancer therapy given for advanced or metastatic disease.
* Not a candidate for definitive therapy (eg, chemoradiation or complete surgical resection).
* Participants with brain metastases are eligible for enrollment, including those with untreated brain metastases. Brain metastases must be asymptomatic and not in need of immediate local therapy. Any untreated brain metastases must be ≤ 20 mm in diameter.
* Any PD-L1 expression (0 to 100%) as determined by VENTANA PD-L1 (SP263) assay, Agilent PD-L1 IHC 22C3 pharmDx, or Agilent PD-L1 IHC 28-8 pharmDx.

Exclusion Criteria:

* Participants with an active autoimmune or inflammatory disease requiring systemic treatment within 2 years.
* Uncontrolled or significant cardiovascular conditions within 6 months prior to enrollment that are ongoing or with risk of recurrence.
* Inadequate bone marrow or liver function or electrocardiogram (ECG) abnormalities.
* Ongoing treatment with concomitant medication known to cause prolonged QTc interval and that cannot be switched to alternative treatment prior to study entry.
* Treatment targeting KRAS G12C mutation (eg, sotorasib, adagrasib) in any setting.
* Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or study drug administration.
* Other protocol-defined Inclusion/Exclusion criteria apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 630 (Estimated)
Dates: Start 2025-04-24 (Actual); Primary Completion 2029-09-07 (Estimated); Study Completion 2032-04-30 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) as Assessed per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 by Blinded Independent Central Review (BICR) | Up to 7 years
Overall Survival (OS) | Up to 7 years

SECONDARY OUTCOMES:
Overall Response (OR) as Assessed per RECIST v1.1 by BICR | Up to 7 years
Duration of Response (DOR) as Assessed per RECIST 1.1 by BICR | Up to 7 years
PFS as Assessed per RECIST v1.1 by Investigator | Up to 7 years
Number of Participants With Adverse Events (AEs) | Up to 90 days from last dose
Number of Participants With Serious Adverse Events (SAEs) | Up to 90 days from last dose
Number of Participants With AEs Leading to Dose Interruption | Up to 90 days from last dose
Number of Participants With AEs Leading to Dose Reduction | Up to 90 days from last dose
Number of Participants With AEs Leading to Treatment Discontinuation | Up to 90 days from last dose
Number of Deaths | Up to 90 days from last dose
Time to Definitive Deterioration by Non-Small Cell Lung Cancer-Symptom Assessment Questionnaire (NSCLC-SAQ) Total Score | Up to 7 years
Change From Baseline in European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-30) Scale/item Score | Up to 90 days from last dose

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (333):
- United States (36):
  - Local Institution - 0347, Birmingham, Alabama
  - Local Institution - 0581, Fullerton, California
  - Local Institution - 0682, Loma Linda, California
  - Local Institution - 0202, Long Beach, California
  - Local Institution - 0623, Santa Barbara, California
  - Local Institution - 0442, Denver, Colorado
  - Local Institution - 0680, Ocala, Florida
  - Local Institution - 0679, Orange City, Florida
  - Local Institution - 0621, Palm Bay, Florida
  - Local Institution - 0377, Tamarac, Florida
  - Local Institution - 0647, Tampa, Florida
  - Local Institution - 0392, Fort Gordon, Georgia
  - Local Institution - 0031, Marietta, Georgia
  - Local Institution - 0665, Arlington Heights, Illinois
  - Local Institution - 0676, Chicago, Illinois
  - Local Institution - 0683, Springfield, Illinois
  - Local Institution - 0684, Fort Wayne, Indiana
  - Local Institution - 0423, Munster, Indiana
  - Local Institution - 0366, Edgewood, Kentucky
  - Local Institution - 0566, Louisville, Kentucky
  - Local Institution - 0644, Shreveport, Louisiana
  - Local Institution - 0385, Columbia, Maryland
  - Local Institution - 0019, Boston, Massachusetts
  - Local Institution - 0437, Worcester, Massachusetts
  - Local Institution - 0293, Detroit, Michigan
  - Local Institution - 0685, Fenton, Missouri
  - Local Institution - 0634, Schenectady, New York
  - Local Institution - 0618, White Plains, New York
  - Local Institution - 0624, Asheville, North Carolina
  - Local Institution - 0672, Salisbury, North Carolina
  - Local Institution - 0688, Easton, Pennsylvania
  - Local Institution - 0657, York, Pennsylvania
  - Local Institution - 0681, Greenville, South Carolina
  - Local Institution - 0658, Greenville, South Carolina
  - Local Institution - 0652, Laredo, Texas
  - Local Institution - 0622, San Antonio, Texas
- Argentina (7):
  - Instituto Alexander Fleming, Ciudad Autónoma de Buenos Aires, Buenos Aires
  - IDIM - Instituto de Investigaciones Metabólicas, Ciudad de Buenos Aires, Buenos Aires
  - Hospital Universitario Austral, Pilar, Buenos Aires
  - Hospital Italiano de Buenos Aires, ABB, Buenos Aires F.D.
  - Local Institution - 0571, Buenos Aires, Buenos Aires F.D.
  - Clinica Adventista Belgrano, CABA, Buenos Aires F.D.
  - Sanatorio Plaza, Rosario, Santa Fe Province
- Australia (9):
  - Canberra Hospital, Canberra, Australian Capital Territory
  - Tamworth Hospital, North Tamworth, New South Wales
  - Orange Hospital, Orange, New South Wales
  - Princess Alexandra Hospital, Brisbane, Queensland
  - Lyell McEwin Hospital, Elizabeth Vale, South Australia
  - Frankston Hospital, Frankston, Victoria
  - Northern Hospital, Melbourne, Victoria
  - Latrobe Regional Health, Traralgon, Victoria
  - Joondalup Health Campus, Joondalup, Western Australia
- Austria (5):
  - Medizinische Universität Graz, Graz, Styria
  - Klinikum Wels-Grieskirchen GmbH, Wels, Upper Austria
  - Kepler Universitätsklinikum, Linz
  - Medizinische Universität Wien, Vienna
  - Local Institution - 0673, Vienna
- Belgium (6):
  - UZ Brussel, Brussels, Bruxelles-Capitale, Région de
  - Cliniques universitaires Saint-Luc, Brussels, Bruxelles-Capitale, Région de
  - Jessa Ziekenhuis, Hasselt, Limburg
  - AZ Maria Middelares, Ghent, Oost-Vlaanderen
  - UZ Leuven, Leuven, Vlaams-Brabant
  - Centre Hospitalier Universitaire de Liège - Domaine Universitaire du Sart Tilman, Liège
- Brazil (15):
  - CEDOES, Vitória, Espírito Santo
  - Nucleo de Oncologia da Bahia, Salvador, Estado de Bahia
  - Cetus Oncologia - Unidade Belo Horizonte, Belo Horizonte, Minas Gerais
  - ONCOSITE - Centro de Pesquisa Clinica em Oncologia, Ijuí, Rio Grande do Sul
  - Hospital São Lucas da PUCRS, Porto Alegre, Rio Grande do Sul
  - Instituto de Oncologia Saint Gallen, Santa Cruz do Sul, Rio Grande do Sul
  - Hospital de Amor Amazônia, Porto Velho, Rondônia
  - Clínica de Oncologia Reichow, Blumenau, Santa Catarina
  - Clínica de Neoplasias Litoral, Itajaí, Santa Catarina
  - Fundação Pio XII - Hospital de Câncer de Barretos, Barretos, São Paulo
  - Advanze Pesquisa, São Carlos, São Paulo
  - Fundação Faculdade Regional de Medicina de São José do Rio Preto, São José do Rio Preto, São Paulo
  - A. C. Camargo Cancer Center, São Paulo, São Paulo
  - Instituto Nacional de Câncer - INCA, Rio de Janeiro
  - Local Institution - 0258, São Paulo
- Bulgaria (4):
  - MBAL Uni Hospital, Panagyurishte, Pazardzhik
  - Multiprofile Hospital for Active Treatment Serdika EOOD, Sofia, Sofia (stolitsa)
  - Complex Oncology Center - Ruse EOOD, Rousse
  - Trakia Hospital, Stara Zagora
- Canada (2):
  - Local Institution - 0074, Halifax, Nova Scotia
  - Local Institution - 0559, Montreal, Quebec
- Chile (2):
  - Bradfordhill, Recoleta, Santiago Metropolitan
  - FALP, Santiago, Santiago Metropolitan
- China (41):
  - The First Afflilated Hospital of Bengbu Medical College, Bengbu, Anhui
  - Anhui Provincial Hospital, Hefei, Anhui
  - Beijing Cancer hospital, Beijing, Beijing Municipality
  - Beijing Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Beijing Chest Hospital,Capital Medical University, Beijing, Beijing Municipality
  - Chongqing University Cancer Hospital, Chongqing, Chongqing Municipality
  - Fujian Medical University Union Hospital, Fuzhou Fujian, Fujian
  - The First Affiliated hospital of Xiamen University, Xiamen, Fujian
  - The First Affiliated Hospital, Sun Yat-sen University, Guangzhou, Guangdong
  - The First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - Cancer Hospital of Shantou University Medical College, Shantou, Guangdong
  - Cancer Hospital Chinese Academy of Medical Sciences. Shenzhen Center, Shenzhen, Guangdong
  - ShenZhen People's Hospital, Shenzhen, Guangdong
  - Guangxi Medical University Affiliated Tumor Hospital, Nanning, Guangxi
  - Fourth Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - Nanyang City Center Hospital, Nanyang, Henan
  - The First Affiliated Hospital of Xinxiang Medical University, Xinxiang, Henan
  - Tongji Hospital Tongji Medical,Science & Technology, Wuhan, Hubei
  - Hunan Cancer Hospital, Changsha, Hunan
  - Nanjing Drum Tower Hospital The Affiliated Hospital of Nanjing University Medical School, Nanjing, Jiangsu
  - The First Affiliated Hospital Of Soochow University, Suzhou, Jiangsu
  - Northern Jiangsu People's Hospital, Yangzhou, Jiangsu
  - The Second Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - The First Hospital of Jilin University, Changchun, Jilin
  - The First Hospital of China Medical University, Shenyang, Liaoning
  - Shengjing Hospital of China Medical University, Shenyang, Liaoning
  - Liaoning Cancer Hospital, Shenyang, Liaoning
  - Shandong Cancer Hospital, Jinan, Shandong
  - LinYi Cancer Hospital, Linyi, Shandong
  - Local Institution - 0470, Shanghai, Shanghai Municipality
  - Local Institution - 0381, Shanghai, Shanghai Municipality
  - Shanghai East Hospital, Shanghai, Shanghai Municipality
  - Shanxi Cancer Hospital, Taiyuan, Shanxi
  - Sichuan Cancer hospital, Chengdu, Sichuan
  - West China Hospital, Sichuan University, Chengdu, Sichuan
  - Tianjin Medical University General Hospital, Tianjin, Tianjin Municipality
  - The first Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Sir Run Run Shaw Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang
  - Taizhou Hospital of Zhejiang Province, Taizhou, Zhejiang
- Colombia (9):
  - Clinica Somer, Rionegro, Antioquia
  - Local Institution - 0191, Puerto Colombia, Atlántico
  - Local Institution - 0189, Bogotá, Bogota D.C.
  - Sociedad De Oncología y Hematología Del Cesar SAS, Valledupar, Cesar Department
  - Instituto Médico de Alta Tecnología S.A.S - IMAT S.A.S, Montería, COR
  - Local Institution - 0671, Bogota, Cundinamarca
  - Fundación Cardiovascular de Colombia, Floridablanca, Santander Department
  - Fundación Valle del Lili, Cali, Valle del Cauca Department
  - Clinica Medellin S.A, Medellín
- Croatia (5):
  - Opća bolnica Dubrovnik, Dubrovnik, Dubrovnik-Neretva County
  - Poliklinika MEDICO - Rijeka, Rijeka, Primorje-Gorski Kotar County
  - Klinički Bolnički Centar Split, Split, Split-Dalmatia County
  - Local Institution - 0567, Osijek
  - Local Institution - 0585, Zagreb
- France (18):
  - Local Institution - 0159, Mulhouse, Alsace
  - Centre François Baclesse, Caen, Calvados
  - Centre Georges François Leclerc, Dijon, Côte-d'Or
  - CHRU de Brest, Brest, Finistère
  - Institut Régional du Cancer Montpellier, Montpellier, Hérault
  - Chu Grenoble Alpes, La Tronche, Isère
  - Local Institution - 0560, Angers, Maine-et-Loire
  - Centre Hospitalier Régional Universitaire de Nancy - Hôpitaux de Brabois, Vandœuvre-lès-Nancy, Meurthe-et-Moselle
  - Institut Paoli-Calmettes, Marseille, Provence-Alpes-Côte d'Azur Region
  - CHU d'Amiens-Picardie - Hôpital Sud, Amiens, Somme
  - Gustave Roussy, Villejuif, Val-de-Marne
  - Hôpital Ambroise Paré, Boulogne-Billancourt
  - Chu Gabriel Montpied, Clermont-Ferrand
  - Centre Hospitalier Universitaire de Limoges - Hôpital Dupuytren, Limoges
  - Assistance Publique Hôpitaux de Marseille - Hôpital Nord, Marseille
  - Local Institution - 0133, Paris
  - Hopitaux Universitaires Paris Centre-Hopital Cochin, Paris
  - Hôpital Nord Guillaume-et-René-Laennec / CHU de Nantes, Saint-Herblain
- Germany (19):
  - Klinikum Esslingen, Esslingen am Neckar, Baden-Wurttemberg
  - Bundeswehrkrankenhaus Ulm, Ulm, Baden-Wurttemberg
  - Klinikum der Ludwig-Maximilians-Universitaet Muenchen, München, Bavaria
  - Centrum für Hämatologie und Onkologie Bethanien, Frankfurt am Main, Hesse
  - UKGM Gießen/Marburg, Giessen, Hesse
  - Praxis Onkologie am Raschplatz, Hanover, Lower Saxony
  - Pius Hospital Oldenburg, Oldenburg, Lower Saxony
  - Klinikum Köln-Merheim, Cologne, North Rhine-Westphalia
  - Evangelisches Krankenhaus Herne - Eickel, Herne, North Rhine-Westphalia
  - Universitätsklinikum Halle, Halle, Saxony-Anhalt
  - Malteser Krankenhaus St. Franziskus-Hospital, Flensburg, Schleswig-Holstein
  - SRH Wald-Klinikum Gera GmbH, Gera, Thuringia
  - Universitätsklinikum Jena, Jena, Thuringia
  - Vivantes Klinikum Neukölln, Berlin
  - Evangelische Lungenklinik Berlin, Berlin
  - Local Institution - 0675, Halle
  - Local Institution - 0528, Hemer
  - Klinikum Stuttgart - Katharinenhospital, Stuttgart
  - Universitaetsklinikum Wuerzburg, Würzburg
- Greece (3):
  - Errikos Dunant Hospital Center, Athens, Attikí
  - Thoracic General Hospital of Athens "I Sotiria", Athens, Attikí
  - University General Hospital of Larissa, Larissa, Thessalía
- Queen Mary Hospital, Hksar, Hong Kong
- Hungary (6):
  - Local Institution - 0144, Gyöngyös - Mátraháza, Heves County
  - Local Institution - 0157, Tatabánya, Komárom-Esztergom
  - Farkasgyepui Tudogyogyintezet, Farkasgyepű, Veszprém megye
  - Semmelweis Egyetem, Budapest
  - Országos Korányi Pulmonológiai Intézet, Budapest
  - Petz Aladar Egyetemi Oktato Korhaz, Győr
- India (15):
  - Local Institution - 0222, Visakhapatnam, Andhra Pradesh
  - Local Institution - 0136, Ahmedabad, Gujarat
  - Local Institution - 0230, Ahmedabad, Gujarat
  - Local Institution - 0155, Thiruvananthapuram, Kerala
  - Local Institution - 0154, Mumbai, Maharashtra
  - Local Institution - 0312, New Delhi, National Capital Territory of Delhi
  - Local Institution - 0511, New Delhi, National Capital Territory of Delhi
  - Local Institution - 0135, New Delhi, National Capital Territory of Delhi
  - Local Institution - 0226, Bhubaneswar, Odisha
  - Local Institution - 0224, Madurai, Tamil Nadu
  - Local Institution - 0663, Hyderabad, Telangana
  - Local Institution - 0153, Varanasi, Uttar Pradesh
  - Local Institution - 0161, Howrah, West Bengal
  - Local Institution - 0221, Kolkata, West Bengal
  - Local Institution - 0661, Hyderabad
- Ireland (5):
  - Cork University Hospital, Cork
  - Mater Private Hospital - Dublin, Dublin
  - St. James's Hospital, Dublin
  - UCD School of Medicine Beacon Hospital, Dublin
  - Beaumont Hospital, Dublin, Dublin
- Israel (5):
  - Rabin Medical Center, Petah Tikva, Central District
  - Sheba Medical Center, Ramat Gan, Central District
  - Yitzhak Shamir Medical Center, Ẕerifin, Central District
  - Hadassah Medical Center, Jerusalem, Jerusalem
  - Carmel Hospital, Haifa, Ḥeifā
- Italy (11):
  - Instituto Tumori Giovanni Paolo II, Bari, Apulia
  - IRCCS - Istituto Romagnolo per lo Studio dei Tumori (IRST) "Dino Amadori", Meldola, Emilia-Romagna
  - A.O.R.N. Ospedale dei Colli - Monaldi V., Naples, Napoli
  - Azienda Ospedaliero-Universitaria San Luigi Gonzaga, Orbassano, Piedmont
  - Istituto Nazionale Tumori Regina Elena, Rome, Roma
  - Azienda Ospedaliera Universitaria Careggi, Florence, Tuscany
  - Ospedale San Martino, Genova
  - Istituto Oncologico Veneto IRCCS, Padua
  - Azienda Ospedaliero Universitaria di Parma, Parma
  - Fondazione IRCCS Policlinico San Matteo, Pavia
  - Local Institution - 0556, Varese
- Japan (25):
  - Local Institution - 0607, Nagoya, Aichi-ken
  - Local Institution - 0305, Nagoya, Aichi-ken
  - Local Institution - 0298, Sapporo, Hokkaido
  - Local Institution - 0304, Kanazawa, Ishikawa-ken
  - Local Institution - 0302, Sagamihara, Kanagawa
  - Local Institution - 0369, Yokohama, Kanagawa
  - Local Institution - 0301, Sendai, Miyagi
  - Local Institution - 0306, Kashihara, Nara
  - Local Institution - 0368, Kurashiki, Okayama-ken
  - Local Institution - 0642, Hirakata, Osaka
  - Local Institution - 0303, Hidaka, Saitama
  - Local Institution - 0300, Ina-machi, Saitama
  - Local Institution - 0606, Hamamatsu, Shizuoka
  - Local Institution - 0299, Shimotsuga, Tochigi
  - Local Institution - 0674, Bunkyo Ku, Tokyo
  - Local Institution - 0343, Toyoma, Toyama
  - Local Institution - 0542, Iwakuni, Yamaguchi
  - Local Institution - 0307, Akashi
  - Local Institution - 0346, Aomori
  - Local Institution - 0310, Fukuoka
  - Local Institution - 0367, Fukushima
  - Local Institution - 0308, Kumamoto
  - Local Institution - 0687, Nagasaki
  - Local Institution - 0297, Osaka
  - Local Institution - 0309, Osaka
- Mexico (9):
  - Local Institution - 0583, Saltillo, Coahuila
  - Local Institution - 0176, Mexico City, DIF
  - Local Institution - 0579, Pachuca, Hidalgo
  - Hospital Civil Fray Antonio Alcalde, Guadalajara, Jalisco
  - Local Institution - 0591, Monterrey, Nuevo León
  - Local Institution - 0175, Chihuahua City
  - Unidad Médica Onco-hematológica, Puebla City
  - Local Institution - 0638, Puebla City
  - Local Institution - 0180, Veracruz
- Netherlands (2):
  - Maastricht UMC+, Maastricht, Limburg
  - Nederlands Kanker Instituut Antoni van Leeuwenhoek (NKI AVL), Amsterdam, North Holland
- Poland (8):
  - Med-Polonia Sp. z o. o., Poznan, Greater Poland Voivodeship
  - Szpital Specjalistyczny im. Henryka Klimontowicza, Gorlice, Lesser Poland Voivodeship
  - Pratia MCM Krakow, Krakow, Lesser Poland Voivodeship
  - Dolnośląskie Centrum Onkologii, Pulmonologii i Hematologii, Wroclaw, Lower Silesian Voivodeship
  - Uniwersytecki Szpital Kliniczny Nr 4 w Lublinie, Lublin, Lublin Voivodeship
  - Centrum Onkologii im. Prof. Franciszka Lukaszczyka, Bydgoszcz
  - Pratia Onkologia Katowice, Katowice
  - Szpital Specjalistyczny w Prabutach Spolka z o.o., Prabuty
- Portugal (3):
  - Instituto Português de Oncologia de Lisboa Francisco Gentil, Lisbon, Lisbon District
  - Instituto Portugês de Oncologia de Coimbra Francisco Gentil, Coimbra
  - Centro Hospitalar do Porto - Hospital de Santo António, Porto
- Romania (12):
  - SC Memorial Healthcare International SRL, Bucharest, București
  - Institutul Oncologic Bucuresti "Prof. Dr. Alexandru Trestioreanu", Bucharest, București
  - Cardiomed SRL Cluj-Napoca, Cluj-Napoca, Cluj
  - SC Radiotherapy Center Cluj SRL, Florești, Cluj
  - Ovidius Clinical Hospital OCH, Ovidiu, Constanța County
  - Centrul de Oncologie "Sfântul Nectarie", Craiova, Dolj
  - Cabinet Medical Oncomed, Timișoara, Timiș County
  - Institutul Oncologic Cluj, Cluj-Napoca
  - Affidea Constanța, Constanța
  - S.C. Centrul de Oncologie Euroclinic S.R.L., Iași
  - Institutul Regional de Oncologie, Iași
  - Spitalul Municipal Schuller Ploiești, Ploieşti
- Saudi Arabia (3):
  - Local Institution - 0614, Jeddah, Makkah Al Mukarramah
  - Local Institution - 0602, Riyadh
  - Local Institution - 0562, Riyadh
- South Korea (8):
  - Chungbuk National University Hospital, Cheongju-si, Chungcheongbuk-do [Chungbuk]
  - Gachon University Gil Medical Center, Namdong-gu, Incheon-gwangyeoksi [Incheon]
  - Pusan National University Yangsan Hospital, Yangsan, Kyǒngsangnam-do
  - Pusan National University Hospital, Busan, Pusan-Kwangyǒkshi
  - Severance Hospital, Yonsei University Health System, Seoul, Seoul-teukbyeolsi [Seoul]
  - Konkuk University Medical Center, Seoul, Seoul-teukbyeolsi [Seoul]
  - Local Institution - 0248, Seoul, Seoul-teukbyeolsi [Seoul]
  - Korea University Guro Hospital, Seoul, Seoul-teukbyeolsi [Seoul]
- Spain (16):
  - CHUAC-Hospital Teresa Herrera, A Coruña, A Coruña [La Coruña]
  - CHUS - Hospital Clinico Universitario, Santiago de Compostela, A Coruña [La Coruña]
  - Hospital Universitari Vall d'Hebron, Barcelona, Barcelona [Barcelona]
  - Local Institution - 0497, Hospitalet, Barcelona [Barcelona]
  - Local Institution - 0505, Barcelona, Catalunya [Cataluña]
  - Hospital Son Llàtzer, Palma, Illes Balears [Islas Baleares]
  - Hospital General Universitario Gregorio Marañon, Madrid, Madrid, Comunidad de
  - Hospital Universitario Ramón y Cajal, Madrid, Madrid, Comunidad de
  - Hospital Universitario 12 de Octubre, Madrid, Madrid, Comunidad de
  - Hospital Universitario Puerta de Hierro Majadahonda, Majadahonda, Madrid, Comunidad de
  - CHUVI- Hospital Alvaro Cunqueiro, Pontevedra, Pontevedra [Pontevedra]
  - Hospital Arnau de Vilanova, Valencia, València
  - Hospital Clinico San Carlos, Madrid
  - H.R.U Málaga - Hospital General, Málaga
  - Hospital Universitario Virgen Del Rocio, Seville
  - Local Institution - 0495, Valencia
- Kantonsspital Münsterlingen - Spital Thurgau AG, Münsterlingen, Switzerland
- Taiwan (5):
  - Chi Mei Hospital - Liouying Branch, Tainan, Tainan
  - Tri-Service General Hospital, Taipei City, Taipei
  - Taipei Medical University Shuang Ho Hospital, New Taipei City
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
- Thailand (3):
  - Chulalongkorn University, Bangkok, Bangkok
  - Faculty of Medicine - Khon Kaen University, Muang, Changwat Khon Kaen
  - Songklanagarind hospital, Hat Yai, Changwat Songkhla
- Turkey (Türkiye) (8):
  - Local Institution - 0199, Izmir, Karsiyaka, İzmir
  - Local Institution - 0197, Adana
  - Hacettepe Universite Hastaneleri, Ankara
  - Ankara University Health Practice and Research Hospitals, Ankara
  - Local Institution - 0198, Ankara
  - Local Institution - 0550, Istanbul
  - TC Saglik Bakanligi Goztepe Prof. Dr. Suleyman Yalcin Sehir Hastanesi, Istanbul
  - Local Institution - 0200, Izmir
- United Kingdom (6):
  - University College London Hospital, London, London, City of
  - Guy's & St Thomas' NHS Foundation Trust, London, London, City of
  - Heartlands Hospital, Birmingham
  - Local Institution - 0545, Guildford
  - The Royal Surrey County Hospital, Guildford
  - Local Institution - 0093, Manchester

IPD SHARING:
Plan to Share IPD: Yes
BMS will provide access to individual anonymized participant data upon request from qualified researchers, and subject to certain criteria. Additional information regarding Bristol Myer Squibb's data sharing policy and process can be found at https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
Supporting Information: Study Protocol, SAP, CSR
Time Frame: See Plan Description
Access Criteria: See Plan Description
URL: https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsclinicaltrials.com/us/en/clinical-trials/NCT06875310.html